CLINICAL TRIAL: NCT04895774
Title: Stool Collection From Healthy Donors for the ex Vivo Study of the Mechanism of Action of Active Ingredients on the Intestinal Microbiota: Bacteria / Host Interaction Model
Brief Title: Ex Vivo Study of the Mechanism of Action of Active Ingredients on the Intestinal Microbiota
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nutri & Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-A00700-41
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Microbial Colonization
MeSH Terms: conditions — Communicable Diseases | interventions — Polyphenols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Probiotic strains — Fresh stools will be cultured in vitro in fermenters with adjunction of probiotic strains
Other: Polyphenols — Fresh stools will be cultured in vitro in fermenters with adjunction of polyphenols
Other: Fibers — Fresh stools will be cultured in vitro in fermenters with adjunction of fibers

SUMMARY:
To design and understand the mechanism of action of different combinations of nutraceuticals coupling bacteria, fibers and polyphenols, which can act on the 4 pillars simultaneously via an innovative ex-vivo model approach coupled with functional and quantitative metagenomics.

DETAILED DESCRIPTION:
The objective of the study is to collect fresh stools from 4 healthy volunteers, in order to study the mechanism of action of probiotic strains, polyphenols and fibers, alone or in combinations. These fresh stools will be cultured in vitro in fermenters, and the samples taken at different culture times will be analyzed in terms of microbial composition (shotgun metagenomic analysis) and their cellular activity (functional metagenomic analysis).

ELIGIBILITY:
Inclusion Criteria:

* Person with a low fiber diet (<17g / day).

Exclusion Criteria:

* Taking antibiotics and / or transit modulators in the 3 months preceding the sample;
* Colonoscopy in the last 3 months;
* Person under legal protection measure (curators, tutors, etc.).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The research will be carried out on 4 healthy volunteers. The research will be carried out by the coordinating team of the INRAE MetaGenoPolis Unit.
Sampling Method: Probability Sample
Enrollment: 4 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Bacterial growth | Day 1 to Day 15
  Change about the bacterial growth after 15 days of incubation
PH evolution | Day 1 to Day 15
  Change about the PH evolution after 15 days of incubation
Quantity of Co2 production | Day 1 to Day 15
  Change about the quantity of Co2 production after 15 days of incubation

IPD SHARING:
Plan to Share IPD: No